CLINICAL TRIAL: NCT04250649
Title: Does Disinfection of the Subcutaneous Tissue Reduce Contamination of the Operating Field With P. Acnes Compared to Dissection With an Electric Cautery During Primary Shoulder Surgery
Brief Title: Does Disinfection of the Subcutaneous Tissue Reduce Contamination of the Operating Field With P. Acnes?
Acronym: Elec_cautery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Hôpital du Valais (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2020-00170
Record Dates: First submitted 2020-01-28; First posted 2020-01-31 (Actual); Last update posted 2020-01-31 (Actual); Status verified 2020-01

CONDITIONS: Surgical Incision
Keywords: subcutaneous desinfection, P. acnes, electric cautery
MeSH Terms: conditions — Surgical Wound

STUDY DESIGN:
Intervention Model Description: This is a single center, category A randomized clinical trial.
Who Masked: Participant, Outcomes Assessor
Masking Description: A standard block randomization strategy will be used. The ratio between intervention and control will be set at 2: 1. This will facilitate recruitment and provide more information on the effectiveness of the intervention. The randomization sequence will be created using the STATA program.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Active Comparator): Betadine solution disinfection of the subcutaneous tissue during primary shoulder surgery
  Interventions: Procedure: subcutaneous tissue disinfection
- Controle (No Intervention): Control group with surgery without disinfection of the subcutaneous tissue but dissection with an electric cautery during primary shoulder surgery

INTERVENTIONS:
Procedure: subcutaneous tissue disinfection — Skin and subcutaneous incision (up to the muscular fascia) with "superficial blade" scalpel, disinfection of the subcutaneous tissue with 3cc of Betadine solution, placement of the retractors, dissection and development of the delto-pectoral interval with "deep blade" scalpel.
  When the joint is opened, bacteriological smears are taken from 5 sites in the two groups. 1) exposed subcutaneous tissue, 2) surgeon's gloves (distal end of fingers), 3) "superficial blade", 4) "deep blade", 5) retractors.
  The rest of the shoulder surgery procedure does not differ from what is commonly performed.
  The samples are sent to bacteriology for bacterial culture. Anaerobic research is done specifically for P. acnes. The results are considered negative after 10 days.
  Arms: Intervention

SUMMARY:
Propionibacterium acnes is a pathogen commonly identified in postoperative shoulder infections. A recent study has shown that P. acnes is likely to be disseminated in the operating field from the subcutaneous layer by the manipulation of soft tissues by the surgeon and the instruments. Disinfection of the subcutaneous tissue seems to significantly reduce contamination of the operating field during primary shoulder surgery. This study seeks to assess the efficacy of disinfection of the subcutaneous tissue compared to dissection with an electrosurgical unit on P. acnes contamination during primary shoulder surgery.

DETAILED DESCRIPTION:
The investigators are going to study the efficacy of disinfecting the subcutaneous tissue with Betadine standard solution during primary shoulder surgery compared to electrosurgical dissection. They will randomize 105 patients on two arms. The control group receiving no disinfection of the subcutaneous tissue but a dissection with an electric cautery(A) and intervention group receiving a disinfection of the subcutaneous tissue (B). They believe that the duration of 4 years is sufficient to recruit the number of patients necessary for this study.

All patients 18 years of age or older admitted to Valais Hospital for primary shoulder surgery and having signed the consent of the study will be eligible.

The use of disinfection of the subcutaneous tissue during primary shoulder surgery could reduce contamination of the operating field and theoretically the post-operative infection rate after primary shoulder surgery.

The study focuses on disinfection with Betadine solution of the subcutaneous tissue during primary shoulder surgery. This action could decrease contamination of the operating field and the infection rate after primary shoulder surgery.

This solution is already widely used for disinfecting the skin and traumatic or surgical wounds.

The investigators will use it according to the recommendations made in the Swiss Compendium of Medicines.

No evidence has been brought to a decrease in this contamination if the dissection is carried out with an electric cautery. Scalpel dissection is used as standard in orthopedic surgery as well as in other surgical disciplines.

ELIGIBILITY:
Inclusion Criteria:

1. = or> 18 years old
2. treated at the Valais Hospital for primary shoulder surgery.
3. have signed the consent

Exclusion Criteria:

1. <18 years old
2. History of shoulder surgery
3. History of shoulder infection
4. Antibiotic therapy in the 2 weeks preceding the intervention
5. Cortisone infiltration in the 6 months preceding the intervention
6. Allergy to iodinated contrast agent or Cefuroxime
7. Allergy to povidone iodine complex or other contraadication to Betadine
8. Refusal of study terms

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 105 (Estimated)
Dates: Start 2020-03-31 (Estimated); Primary Completion 2022-03-31 (Estimated); Study Completion 2024-03-31 (Estimated)

PRIMARY OUTCOMES:
positive sample | 4 years
  Compare the positive bacteriological sample rate during an open shoulder surgery procedure with a disinfection of the subcutaneous tissue compared to an operating procedure without disinfection but dissection with an electric knife.

CONTACTS AND LOCATIONS:
Overall Officials: Beat K Moor, PD Dr, Principal Investigator — Hopital du Valais
Locations (1):
- Hôpital du Valais, Martigny-Ville, Valais, Switzerland

IPD SHARING:
Plan to Share IPD: No